CLINICAL TRIAL: NCT05974995
Title: Robotic-assisted Versus Conventional Laparoscopic Surgery in the Management of Obese Patients With Early Endometrial Cancer in the Sentinel Lymph Node Era: a Randomized Controlled Study
Brief Title: Robotic-assisted Versus Conventional Laparoscopic Surgery in Obese Patients With Early Endometrial Cancer
Acronym: RObese
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Fanfani Francesco, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5798
Record Dates: First submitted 2023-07-18; First posted 2023-08-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Endometrial Cancer; Endometrial Neoplasms; Obesity, Morbid; Gynecologic Cancer; Gynecologic Disease
MeSH Terms: conditions — Endometrial Neoplasms; Obesity, Morbid; Genital Diseases, Female | interventions — Robotic Surgical Procedures; Laparoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic surgery (Experimental)
  Interventions: Procedure: Robot-assisted surgery
- Laparoscopic surgery (Active Comparator)
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Robot-assisted surgery — Total hysterectomy with bilateral salpingo-oophorectomy and lymphnodes staging using DaVinci Xi
  Arms: Robotic surgery
Procedure: Laparoscopic surgery — Total hysterectomy with bilateral salpingo-oophorectomy and lymph nodes staging using standard laparoscopic approach
  Arms: Laparoscopic surgery

SUMMARY:
Data across literature suggest that robotic surgery may offer benefit specifically in patient with morbid obesity with endometrial cancer, but to date no randomized trials have been conducted to confirm these observations.

This randomized controlled multicentric trial aims to evaluate the most appropriate minimally invasive surgical approach in morbidly obese (BMI >= 30) patients with endometrial carcinoma.

DETAILED DESCRIPTION:
Background:

Endometrial cancer is the fourth cancer in women, the most common gynecologic cancer in high-income countries and the second most common gynecologic cancer worldwide.

The high incidence of endometrial cancer is associated with several risk factors, but the growing prevalence of obesity has been identified as one of the majors. Many patients with endometrial cancer are obese and have clinically relevant coexisting conditions that negatively affects anesthesiological parameters and surgical performance when patients undergo surgery, thus potentially increasing the risk of peri-operative complications.

For patients presenting at early-stage disease the standard procedure is total hysterectomy with bilateral salpingo-oophorectomy and lymph nodal staging. Prospective and retrospective studies demonstrate that compared to systemic lymphadenectomy, sentinel lymph node mapping have high accuracy in detecting nodal metastases, and together with ultrastaging may increase the detection of lymph node metastasis with low false-negative rates in patients with apparent uterine-confined disease. Also, recent evidence proved sentinel lymph node biopsy to be a feasible and safe alternative to lymphadenectomy in high-risk endometrial cancer.

Many randomized prospective studies proved laparoscopic surgical staging to be feasible in terms of short-term outcomes, equivalent in disease-free survival and no different in overall survival, thus the current surgical approach is minimally invasive. Also, innovative surgical approaches such as robotic surgery have been exploited showing equivalent oncologic outcomes when compared to traditional laparoscopic surgery.

In 2015, Uccella et al. proved that laparoscopy is superior to open surgery even in case of morbid obesity. Particularly, minimally invasive surgery has been shown to have faster recovery and a higher likelihood of retroperitoneal staging in morbid obese patients, even if the number of women who received lymphadenectomy was found to be stable up to class II of obesity and then dramatically decreased to 30% for BMI>40. Similarly, the number of lymph nodes removed (when lymphadenectomy was accomplished), decreased significantly in class III obesity. However, the removal of lymph nodes can be less relevant in the era of sentinel lymph node. Once, the completing of lymphadenectomy could imply the need of conversion. In fact, the Gynecologic Oncology Group LAP2 trial showed that the odds of conversion to laparotomy during laparoscopic staging increased significantly with each unit increase in BMI, but the reason for conversion was mainly when an adequate surgical staging cannot be completed.

In many retrospective studies robotic surgery has been shown to have advantages when compared to laparoscopy in obese patients. Cusimano et al published a systematic review and meta-analysis aiming to evaluate rates of conversion to laparotomy with laparoscopy or robotic surgery specifically in patients with endometrial cancer and BMI >30Kg/m2: they included 51 observational studies with a total of 10,800 patients overall and found out that although the conversion rate for patients with BMI>30 Kg/m2 is comparable between laparoscopy and robotic surgery, the proportion of patients with BMI >40 kg/m2 who experienced conversion seems to be higher in laparoscopy compared with robotic. Different reasons were described for conversion: organ/vessel injury, uterine size, advanced/ metastatic disease, inadequate exposure because of adhesions or visceral adiposity, anesthesiologic indications.

In conclusion, data across literature suggest that robotic surgery may offer benefit specifically in patient with morbid obesity, but to date no randomized trials have been conducted to confirm these observations. Furthermore, conclusive data are needed to evaluate length of hospitalization, intraoperative and postoperative complications, adherence to the MSKCC nodal staging algorithm, and oncological outcomes in this group of patients. Robust data in morbidly obese endometrial cancer patients to choose the most appropriate surgical technique are missing, particularly in the era of sentinel lymph node. Moreover, conversion to laparotomy in the previous study occurred to achieve a complete surgical staging with lymphadenectomy. Thus, investigators expect to have a lower conversion rate in this study.

Rationale:

The rationale of the study is to find the most appropriate minimally invasive surgical approach in morbidly obese patients with endometrial carcinoma

Objectives:

Primary objective: To evaluate conversion rate to laparotomy with robotic surgery vs laparoscopic surgery (laparoscopic surgery referent group)

Secondary objectives:

* To evaluate difference in overall duration of surgery
* To evaluate difference in perioperative complications
* To evaluate the adherence to sentinel lymph node MSKCC algorithm
* To compare ergonomics of the two different surgical approach
* To compare quality of life (QoL) at baseline, 1 and 4 weeks (early), and 3 and 6 months (late) after surgery, using the Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire
* To assess adherence to ESGO surgical Quality Index (QI, rate of uterine rupture)
* To evaluate difference in overall survival and disease-free survival

Primary end point: the number of surgical procedures that need a conversion over the total number of surgical procedures in the two arms.

Secondary end points:

* Duration in minutes of surgery
* Number of patients with at least one perioperative complications measured by Clavien Dindo
* To evaluate the ergonomics through the Rapid Upper Limb Assessment (RULA) assessment tool
* Disease-Free Survival (DFS) defined as the time between randomization and the first detection of relapse or death, whichever event occurs first; for patients without events DFS will be censored at the date of last follow-up
* Overall Survival (OS) defined as the time between randomization and death for any cause; for alive patients OS will be censored at the date of last follow-up

Study Design: Randomized Controlled Multicentric Superiority trial

ELIGIBILITY:
Inclusion Criteria:

* BMI >=30
* Age > 18
* Histologically confirmed endometrioid endometrial cancer
* Clinical early stage (stage I)
* No contraindication for minimally invasive surgery
* ASA<4
* Written informed consent.

Exclusion Criteria:

* High probability of laparotomy related to uterine volume (US estimated weight >250 g)
* Concomitant pelvic disease, or anatomical characteristics of the patient
* (Use of uterine manipulator)
* Age >75 years

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | At the end of the enrollment phase
  Number of procedures converted to laparotomy from MIS

SECONDARY OUTCOMES:
Difference in overall duration of surgery | At the end of the enrollment phase
  Difference in duration of procedures measured in minutes
Difference in perioperative complications | 36 and 72 months
  Number of patients with at least one perioperative complications measured by Clavien Dindo
Adherence to sentinel lymph node MSKCC algorithm | At the end of the enrollment phase
  Number of case with completed lymph nodal staging according to MSKCC algorithm
Ergonomics of the two different surgical approach | At the end of the enrollment phase
  Investigators will evaluate the ergonomics of the two MIS system through the Rapid Upper Limb Assessment (RULA) assessment tool. Rula is aimed to make a rapid assessment on neck and upper limb loading in tasks. The risk of work-related disorders is calculated into a score of 1(low) to 7 (high)
Quality of life (QoL) at baseline, 1 and 4 weeks (early), and 3 and 6 months (late) after surgery | 1 and 4 weeks (early), and 3 and 6 months (late) after surgery
  Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire will be used. The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire designed to measure physical, social, emotional, and functional well-being in cancer patients. The score range 0-108; the higher the score, the better the QOL.
Adherence to ESGO surgical Quality Index | 36 and 72 months
  Investigators will assess adherence to ESGO surgical Quality Index (QI, rate of uterine rupture)
Difference in overall survival and disease-free survival | 36 and 72 months
  Investigators will evaluate difference in Overall Survival, defined as the time between randomization and death for any cause, for alive patients OS will be censored at the date of last follow-up; investigators will evaluate difference in disease-free survival, defined as the time between randomization and the first detection of relapse or death, whichever event occurs first; for patients without events DFS will be censored at the date of last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Fanfani, MD, Principal Investigator — Policlinico Gemelli IRCCS
Locations (1):
- Policlinico Gemelli IRCCS, Rome, Italy

REFERENCES:
- [Derived] Dinoi G, Tarantino V, Bizzarri N, Perrone E, Capasso I, Giannarelli D, Querleu D, Giuliano MC, Fagotti A, Scambia G, Fanfani F. Robotic-assisted versus conventional laparoscopic surgery in the management of obese patients with early endometrial cancer in the sentinel lymph node era: a randomized controlled study (RObese). Int J Gynecol Cancer. 2024 May 6;34(5):773-776. doi: 10.1136/ijgc-2023-005197. PMID 38326228

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT05974995/Prot_SAP_001.pdf